CLINICAL TRIAL: NCT04526431
Title: Tacrolimus Pharmacokinetic Subpopulations: Prospective Mechanistic Investigations of the Tacrolimus C/D Ratio
Brief Title: Tacrolimus Pharmacokinetic Subpopulations
Acronym: TIPS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Chiesi SA/NV (Other)
Responsible Party: Sponsor
Other Study IDs: TIPS
Record Dates: First submitted 2020-07-21; First posted 2020-08-25 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Kidney Transplant Failure and Rejection; Immunosuppression-related Infectious Disease
Keywords: Kidney transplantation; Pharmacokinetic; Tacrolimus; Concentration-dose ratio; Pharmacogenetic
MeSH Terms: conditions — Rejection, Psychology | interventions — Dosage Forms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The main result of the TIPS study will be longitudinal trough concentrations of tacrolimus metabolites, over the four first years post-transplantation.
  In order to explain the tacrolimus C/D ratio differences, confounding factors will also be investigated, such as CYP3A4, CYP3A4 and ABCB1 genotypes. DNA will therefore be sampled on the day of inclusion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Tacrolimus once-daily: Patients receiving tacrolimus as a once-daily formulation (Envarsus)
  Interventions: Drug: Dosage Forms Oral
- Tacrolimus bid: Patients receiving tacrolimus as a twice-a-day formulation.
  Interventions: Drug: Dosage Forms Oral

INTERVENTIONS:
Drug: Dosage Forms Oral — Dosage form of tacrolimus (extended release tacrolimus or immediate release tacrolimus)

SUMMARY:
This prospective study will investigate the concentrations of tacrolimus metabolites (M-I and M-III) over the four first years post-transplantation.

A differential metabolism might result in different metabolites' concentration and explain a kidney survival difference between "high rate metabolism" (defined as a concentration/dose ratio, C/D ratio, lower than 1.04 µg/l/mg) and other patients.

The primary endpoint is therefore to compare tacrolimus metabolites' concentrations with respect to the group, either < or >= 1.04 µg/l/mg, in order to detect differences in tacrolimus metabolization between these groups.

DETAILED DESCRIPTION:
Tacrolimus is the cornerstone of immunosuppression in renal transplantation, but its nephrotoxicity, in particular, makes it a drug with a narrow therapeutic range, requiring regular pharmacokinetic monitoring. Several studies have demonstrated a relationship between concentration (residual tacrolimus) and dose (prescribed daily tacrolimus) ratio, or C/D ratio, and graft survival. "Fast metabolizers" have been identified by a C/D ratio of less than 1.05 and have poorer graft survival than other renal transplant recipients. The determinants of the C/D ratio (the clinical or biological factors influencing the C/D ratio) are not known.

The purpose of the TIPS study is to prospectively identify tacrolimus metabolism patterns, based on the C/D ratio, and to identify the determinants of the C/D ratio.

The investigators assumed that different metabolism profiles are associated with different degradation profiles of tacrolimus. These degradation profiles can be identified by analysis of known plasma metabolites of tacrolimus (M-I and M-III) and by pharmacogenetic analysis of genes involved in the metabolism of tacrolimus. Also, since the pharmacokinetic profile can be associated with the therapeutic strategy (prolonged-release vs. immediate-release tacrolimus form), it will be investigated in the study in parallel. The hypothesis of this work is that the pharmacokinetic parameters of tacrolimus and its metabolites are associated with renal transplant survival and simultaneously with the therapeutic strategy of the drug. The investigators hope that this will explain the relationship between the C/D ratio of tacrolimus and graft survival, in order to tailor tacrolimus treatment to individual patients (adaptation of the therapeutic strategy, choice of optimal dose).

For this prospective tri-centric randomized prospective study, new renal transplant patients who are scheduled to receive immunosuppression including tacrolimus will be included and randomized between two therapeutic strategies (prolonged-release vs. immediate-release tacrolimus form) within 7 days after transplantation. Patients will be followed for 4 years. Regular consultations will be provided (W6, M3, M6, M12, M24, M36 and M48) including usual biological analyses for renal transplant follow-up, full prescriptions and adherence questionnaire (BAASIS) but also a systematic biopsy of the renal transplant (M3 and M12) and an abbreviated pharmacokinetic study of tacrolimus exposure (M3).

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant patients at the CHUGA, CHU Saint-Etienne or CHU Clermont-Ferrand, whose new transplant is no more than 7 days old (inclusive)
* Patients initially treated with tacrolimus as an immunosuppressant, combined with mycophenolate (MMF), mycophenolic acid (MPA) or everolimus (EVR), with or without corticotherapy.
* No plans to remove tacrolimus from the patient's immunosuppressive treatment (e.g. no plans to switch to belatacept a priori), during the first 4 years post-transplantation.
* Affiliation to or beneficiary of a social security scheme
* Able to read and understand the terms of the protocol
* Informed consent obtained, including specific consent for genetic analysis of target genes.
* For women of childbearing potential, presence of effective contraception (already acquired for patients treated with mycophenolic acid as an immunosuppressant).

Exclusion Criteria:

* Contraindication to the use of tacrolimus
* Patient already treated with tacrolimus at the time of transplantation
* Pregnant, parturient or breastfeeding women
* Patient deprived of liberty by judicial or administrative decision
* Patient under guardianship or curatorship, or receiving forced psychiatric care
* Person admitted to a health or social institution
* Subject cannot be contacted in case of emergency
* Subject in period of exclusion from another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is made of kidney transplant patients with living or deceased donors at Grenoble University Hospital, Saint Etienne University Hospital or Clermont-Ferrand University Hospital.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2020-07-28 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Tacrolimus metabolite concentration | month 3
  The concentration of tacrolimus metabolites M-I and M-III will be evaluated by liquid chromatography / tandem mass spectrometry (LC-MS/MS) given in micrograms per litre (μg/l).
Genotyping | Enrollment
  Genotypes of target genes involved in tacrolimus metabolism (CYP450 3A5, CYP450 3A4, ABCB1)
Tacrolimus residual concentration | month 3
  In addition to the Tacrolimus residual concentration assessed at each visit, this measure will also be performed at T0, T+1h and T+3h for immediate-release tacrolimus and T0, T+1h and T+8h for prolonged-release tacrolimus after treatment. The measurement at T+8h will be carried out on blotting paper with a drop of capillary blood which will be returned by mail, using an envelope given to the patient during the visit. These three measuring points will be used to identify the abbreviated kinetics of tacrolimus during M3 visit.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas JOUVE, MD, PhD, Principal Investigator — University Hospital, Grenoble; Lionel ROSTAING, MD, PhD, Study Chair — University Hospital, Grenoble
Locations (2):
- France (2):
  - Grenoble University Hospital, Grenoble, Auvergne-Rhône-Alpes
  - Saint Etienne University Hospital, Saint-Etienne, Auvergne-Rhône-Alpes

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jouve T, Fonrose X, Noble J, Janbon B, Fiard G, Malvezzi P, Stanke-Labesque F, Rostaing L. The TOMATO Study (Tacrolimus Metabolization in Kidney Transplantation): Impact of the Concentration-Dose Ratio on Death-censored Graft Survival. Transplantation. 2020 Jun;104(6):1263-1271. doi: 10.1097/TP.0000000000002920. PMID 31415035
- [Background] Jouve T, Noble J, Rostaing L, Malvezzi P. An update on the safety of tacrolimus in kidney transplant recipients, with a focus on tacrolimus minimization. Expert Opin Drug Saf. 2019 Apr;18(4):285-294. doi: 10.1080/14740338.2019.1599858. Epub 2019 Apr 1. PMID 30909754
- [Background] Tholking G, Fortmann C, Koch R, Gerth HU, Pabst D, Pavenstadt H, Kabar I, Husing A, Wolters H, Reuter S, Suwelack B. The tacrolimus metabolism rate influences renal function after kidney transplantation. PLoS One. 2014 Oct 23;9(10):e111128. doi: 10.1371/journal.pone.0111128. eCollection 2014. PMID 25340655
- [Background] Egeland EJ, Robertsen I, Hermann M, Midtvedt K, Storset E, Gustavsen MT, Reisaeter AV, Klaasen R, Bergan S, Holdaas H, Hartmann A, Asberg A. High Tacrolimus Clearance Is a Risk Factor for Acute Rejection in the Early Phase After Renal Transplantation. Transplantation. 2017 Aug;101(8):e273-e279. doi: 10.1097/TP.0000000000001796. PMID 28452920